CLINICAL TRIAL: NCT03240731
Title: Bone Marrow Transplantation HLA Haploidentical After a Reduced Intensity Conditioning and Prevention of GvHD Based on Post-transplant Cyclophosphamide Administration in Patients With Severe Sickle Cell Disease
Brief Title: HLA Haploidentical Bone Marrow Transplant in Patients With Severe Sickle Cell Disease
Acronym: DREPHAPLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Keocyt (Unknown); Association Clinique Thérapeutique Infantile du val de Marne (Other)
Responsible Party: Principal Investigator, Nathalie Dhédin, Principal Investigator, Saint-Louis Hospital, Paris, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DREPHAPLO
Record Dates: First submitted 2017-07-31; First posted 2017-08-07 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; haploidentical; graft; marrow
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Bone Marrow Transplantation

STUDY DESIGN:
Intervention Model Description: Haploidentical Marrow Transplants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- bone marrow transplant (Experimental): All the included patient will receive an haploidentical bone marrow transplant with the following protocol concerning the conditioning and GvHD prevention
  Conditioning
  * THYMOGLOBULINE : 0.5mg/kg at D-9 and 2 mg/kg at D-8 and D-7
  * THIOTEPA: 10mg/kg/j at D-7
  * CYCLOPHOSPHAMIDE (Endoxan®):14.5mg/kg/j at D-6 and D-5
  * FLUDARABINE (Fludara®): 30mg/m2 per Day from D-6 to D-2
  * TBI : 2GY : D -1 Graft : Injection at D0 of G-CSF-stimulated bone marrow transplant.
  Prophylaxis of GvHD
  * CYCLOPHOSPHAMIDE (Endoxan®): 50mg/Kg per Day from D+3 to D+4
  * Sirolimus and MycophénolateMofétil (MMP) from D+5. In the absence of acute GvHD (aGvHD), stop of MMP to D35 and pursuit of sirolimus 1 year after the graft.
  Interventions: Biological: bone marrow transplant

INTERVENTIONS:
Biological: bone marrow transplant — haploidentical bone marrow transplant

SUMMARY:
multicentric interventional biomedical research phase II, prospective, non-randomized evaluating a haploidentical marrow transplants after reduced-intensity conditioning and prevention of GvHD based on cyclophosphamide administration post transplantation in patients with severe sickle cell disease.

DETAILED DESCRIPTION:
Sickle cell disease is a severe disease with frequent occurrence of painful crises and progressive installation of a multi organ injuries. Despite the progress in its management, particularly since the introduction of hydroxycarbamide, the median age of death in sickle cell patients was about 40 years in a recent US study. Severe forms resistant to hydroxyurea or cerebral vasculopathy require transfusion programs throughout susceptible to risks of iron overload and alloimmunization. The bone marrow transplantation cures almost 95% of children and adolescents transplant from an HLA-identical siblings. In patients without HLA-identical donor, interesting results have been reported in haploidentical transplants marrow without ex vivo T cell depletion taken after non myeloablative conditioning regimen and GvHD prevention with cyclophosphamide high dose injection after bone marrow transplant . This approach performed in 14 patients was effective to cure 50% of the patients and 50% have rejected the transplant . No death or severe GvHD were related to the procedure.

DREPHAPLO protocol aims to evaluate that approach in a population of sickle cell patients with severe complications of the disease, bringing direct benefit to patients with a cure of the disease in at least half of them.

ELIGIBILITY:
Inclusion criteria recipient:

* Age: 13 years-40 years
* Severe Sickle cell with at least one of the following criteria:

  * Stenosing vasculopathy with abnormal MRA despite prolonged transfusion program
  * PAH confirmed by right catheterization with mPAP> 25mmHg
  * Systolic ejection fraction <55% and tricuspid regurgitation speed> 2.5m /s at distance from an acute episode
  * No possibility of blood transfusion or very complicated blood transfusion
  * Report albumin / creatinine> 30 mg / mmol, confirmed 3 times, away at distance from acute episode and persistent despite hydroxyurea or IEC
  * GFR <80ml / min /1.73m2 (CKD-Epi without ethnic criterion)
  * Previous history of acute liver sequestration with liver failure
  * Acute chest syndrome or vaso-occlusive crises under hydroxyurea
  * Complications of sickle cell transfusion imposing an exchange program with no possible withdrawal beyond a period of one year
* Not having geno-identical donor, but a haploidentical major donor (parent, sibling, adult child, or HbAA AS)
* Having red and understood the information letter and signed the informed consent
* Patients affiliated to a social security system (Social Security or Universal Medical Coverage)

Exclusion Criteria recipient:

* Patient with a geno-identical donor
* Performans status: ECOG> 1
* lung disease: FEV1 and FVC <50% predicted,
* score of PAH NYHA≥2
* Liver disease with bilirubin> 50 .mu.mol / L
* heart failure defined by NYHA≥3 score ejection fraction <45% or shortening fraction <24%
* anti HLA alloimmunization against the donor or against red cell antigens of the donor
* Serology or HIV viral load positively
* Patients who for family, social or geographical reasons, do not wish to be regularly monitored in consultation
* severe uncontrolled infection at the time of inclusion or graft
* pregnant woman (positive beta HCG) or during lactation
* incapable adult patient, trust, guardianship, or safeguard justice

Inclusion criteria donor

* Age> 18 years and <60 years
* Viral serologic economy allows the graft
* No contraindication for general anesthesia
* No contraindication the administration of G-CSF (the existence of sickle cell trait is not a contraindication)
* Lack antigens HLA recognized by the recipient antibody
* Hemoglobin S <50%
* When several donors are compatible: choose according to the ABO recipient: prefer ABO compatibility and major incompatibility and minor incompatibility, and finally major and minor incompatibility.
* Signature of informed consent
* Non-inclusion criteria donors: β HCG positive or known pregnancy

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Survival rate | 2 years
  Survival without sickle cell survival rate (electrophoresis of hemoglobin similar to that from the donor, that is to say a percentage of HbS not exceeding 10% of that of distance donor transfusions and that of a stable manner and without GvHDc other than mild

SECONDARY OUTCOMES:
Survival rate | 1 year
  Survival without sickle cell survival rate (electrophoresis of hemoglobin similar to that from the donor, that is to say a percentage of HbS not exceeding 10% of that of distance donor transfusions and that of a stable manner and without GvHDc other than mild
haematologic reconstitution | 2 years
  defined as a neutrophil count> 500 / mm3 and platelets> 20000 / mm3, for three consecutive days.
Chimerism | at month 1
  Chimerism in the peripheral blood of the total population and the CD3 + population with the techniques usually employed by the centers
Chimerism | at month 2
  Chimerism in the peripheral blood of the total population and the CD3 + population with the techniques usually employed by the centers
Chimerism | at month 3
  Chimerism in the peripheral blood of the total population and the CD3 + population with the techniques usually employed by the centers
Chimerism | at month 4
  Chimerism in the peripheral blood of the total population and the CD3 + population with the techniques usually employed by the centers
Chimerism | at month 5
  Chimerism in the peripheral blood of the total population and the CD3 + population with the techniques usually employed by the centers
Chimerism | at month 6
  Chimerism in the peripheral blood of the total population and the CD3 + population with the techniques usually employed by the centers
Chimerism | at month 9
  Chimerism in the peripheral blood of the total population and the CD3 + population with the techniques usually employed by the centers
Chimerism | at month 12
  Chimerism in the peripheral blood of the total population and the CD3 + population with the techniques usually employed by the centers
Chimerism | at month 24
  Chimerism in the peripheral blood of the total population and the CD3 + population with the techniques usually employed by the centers
hemoglobin electrophoresis | at 1 month
hemoglobin electrophoresis | at 2 month
hemoglobin electrophoresis | at 3 months
hemoglobin electrophoresis | at 4 months
hemoglobin electrophoresis | at 5 months
hemoglobin electrophoresis | at 6 months
hemoglobin electrophoresis | at 9 months
hemoglobin electrophoresis | at 12 months
hemoglobin electrophoresis | at 24 months
occurence of graft versus host disease | at month 24
  evaluated monthly from M1 to M6, and M9, M12, M24
grade of graft versus host disease | at month 24
  Incidence and grade of GvHD, toxic deaths and infectious complications and secondary cancer
occurrence of toxic deaths | at month 24
occurrence of infectious complications | at month 24
occurrence of secondary cancer | at month 24
Lymphocyte immunophenotyping | 2 years
  Lymphocyte immunophenotyping T, B and NK + The Extended Phenotype including activation markers, assessment of naive people and memories, T reg populations etc) and plasma protein electrophoresis: 1 month, 3 months, 6 months, 12 months and 24 months post-transplantation.
ECOG score value | 2 years
  Index Trading ECOG complete physical examination with determination of weight
Assessment of sickle cell disease complications | at 1 year
  Microalbuminuria, creatinuria; echocardiography for measurement of systolic ventricular ejection fraction (February), PAH research and measurement IT Vmax; respiratory function tests with measurement of DLCO; MRI brain with ARM and Cervical Pre-transplant anomalies; Radio of the pelvis
ferritin dosage | at month 3
  Evaluation of iron overload by ferritin
ferritin dosage | at month 6
  Evaluation of iron overload by ferritin
MRI iron overload | at 12 months
  hepatic and cardiac MRI to assess the iron overload

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU Henri-Mondor, Créteil
  - intercommunal hospital of Créteil, Créteil
  - CHU La Timone, Marseille
  - Hospital Necker, Paris
  - Hospital Robert-Debré, Paris
  - Saint-Louis hospital, Paris
  - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yawn BP, Buchanan GR, Afenyi-Annan AN, Ballas SK, Hassell KL, James AH, Jordan L, Lanzkron SM, Lottenberg R, Savage WJ, Tanabe PJ, Ware RE, Murad MH, Goldsmith JC, Ortiz E, Fulwood R, Horton A, John-Sowah J. Management of sickle cell disease: summary of the 2014 evidence-based report by expert panel members. JAMA. 2014 Sep 10;312(10):1033-48. doi: 10.1001/jama.2014.10517. PMID 25203083
- [Background] Habibi A, Arlet JB, Stankovic K, Gellen-Dautremer J, Ribeil JA, Bartolucci P, Lionnet F; centre de reference maladies rares << syndromes drepanocytaires majeurs >>. [French guidelines for the management of adult sickle cell disease: 2015 update]. Rev Med Interne. 2015 May 11;36(5 Suppl 1):5S3-84. doi: 10.1016/S0248-8663(15)60002-9. French. PMID 26007619
- [Background] Lanzkron S, Carroll CP, Haywood C Jr. Mortality rates and age at death from sickle cell disease: U.S., 1979-2005. Public Health Rep. 2013 Mar-Apr;128(2):110-6. doi: 10.1177/003335491312800206. PMID 23450875
- [Background] Bernaudin F, Socie G, Kuentz M, Chevret S, Duval M, Bertrand Y, Vannier JP, Yakouben K, Thuret I, Bordigoni P, Fischer A, Lutz P, Stephan JL, Dhedin N, Plouvier E, Margueritte G, Bories D, Verlhac S, Esperou H, Coic L, Vernant JP, Gluckman E; SFGM-TC. Long-term results of related myeloablative stem-cell transplantation to cure sickle cell disease. Blood. 2007 Oct 1;110(7):2749-56. doi: 10.1182/blood-2007-03-079665. Epub 2007 Jul 2. PMID 17606762
- [Background] Kuentz M, Robin M, Dhedin N, Hicheri Y, Peffault de Latour R, Rohrlich P, Bordigoni P, Bruno B, Socie G, Bernaudin F. Is there still a place for myeloablative regimen to transplant young adults with sickle cell disease? Blood. 2011 Oct 20;118(16):4491-2; author reply 4492-3. doi: 10.1182/blood-2011-07-367490. No abstract available. PMID 22021455
- [Background] Angelucci E, Matthes-Martin S, Baronciani D, Bernaudin F, Bonanomi S, Cappellini MD, Dalle JH, Di Bartolomeo P, de Heredia CD, Dickerhoff R, Giardini C, Gluckman E, Hussein AA, Kamani N, Minkov M, Locatelli F, Rocha V, Sedlacek P, Smiers F, Thuret I, Yaniv I, Cavazzana M, Peters C; EBMT Inborn Error and EBMT Paediatric Working Parties. Hematopoietic stem cell transplantation in thalassemia major and sickle cell disease: indications and management recommendations from an international expert panel. Haematologica. 2014 May;99(5):811-20. doi: 10.3324/haematol.2013.099747. PMID 24790059
- [Background] Hsieh MM, Fitzhugh CD, Weitzel RP, Link ME, Coles WA, Zhao X, Rodgers GP, Powell JD, Tisdale JF. Nonmyeloablative HLA-matched sibling allogeneic hematopoietic stem cell transplantation for severe sickle cell phenotype. JAMA. 2014 Jul 2;312(1):48-56. doi: 10.1001/jama.2014.7192. PMID 25058217
- [Background] Bolanos-Meade J, Fuchs EJ, Luznik L, Lanzkron SM, Gamper CJ, Jones RJ, Brodsky RA. HLA-haploidentical bone marrow transplantation with posttransplant cyclophosphamide expands the donor pool for patients with sickle cell disease. Blood. 2012 Nov 22;120(22):4285-91. doi: 10.1182/blood-2012-07-438408. Epub 2012 Sep 6. PMID 22955919
- [Background] Kamani NR, Walters MC, Carter S, Aquino V, Brochstein JA, Chaudhury S, Eapen M, Freed BM, Grimley M, Levine JE, Logan B, Moore T, Panepinto J, Parikh S, Pulsipher MA, Sande J, Schultz KR, Spellman S, Shenoy S. Unrelated donor cord blood transplantation for children with severe sickle cell disease: results of one cohort from the phase II study from the Blood and Marrow Transplant Clinical Trials Network (BMT CTN). Biol Blood Marrow Transplant. 2012 Aug;18(8):1265-72. doi: 10.1016/j.bbmt.2012.01.019. Epub 2012 Feb 16. PMID 22343376
- [Background] Luznik L, O'Donnell PV, Symons HJ, Chen AR, Leffell MS, Zahurak M, Gooley TA, Piantadosi S, Kaup M, Ambinder RF, Huff CA, Matsui W, Bolanos-Meade J, Borrello I, Powell JD, Harrington E, Warnock S, Flowers M, Brodsky RA, Sandmaier BM, Storb RF, Jones RJ, Fuchs EJ. HLA-haploidentical bone marrow transplantation for hematologic malignancies using nonmyeloablative conditioning and high-dose, posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2008 Jun;14(6):641-50. doi: 10.1016/j.bbmt.2008.03.005. PMID 18489989
- [Background] McCurdy SR, Kanakry JA, Showel MM, Tsai HL, Bolanos-Meade J, Rosner GL, Kanakry CG, Perica K, Symons HJ, Brodsky RA, Gladstone DE, Huff CA, Pratz KW, Prince GT, Dezern AE, Gojo I, Matsui WH, Borrello I, McDevitt MA, Swinnen LJ, Smith BD, Levis MJ, Ambinder RF, Luznik L, Jones RJ, Fuchs EJ, Kasamon YL. Risk-stratified outcomes of nonmyeloablative HLA-haploidentical BMT with high-dose posttransplantation cyclophosphamide. Blood. 2015 May 7;125(19):3024-31. doi: 10.1182/blood-2015-01-623991. Epub 2015 Mar 26. PMID 25814532
- [Background] Bashey A, Zhang X, Sizemore CA, Manion K, Brown S, Holland HK, Morris LE, Solomon SR. T-cell-replete HLA-haploidentical hematopoietic transplantation for hematologic malignancies using post-transplantation cyclophosphamide results in outcomes equivalent to those of contemporaneous HLA-matched related and unrelated donor transplantation. J Clin Oncol. 2013 Apr 1;31(10):1310-6. doi: 10.1200/JCO.2012.44.3523. Epub 2013 Feb 19. PMID 23423745
- [Background] Bashey A, Zhang X, Jackson K, Brown S, Ridgeway M, Solh M, Morris LE, Holland HK, Solomon SR. Comparison of Outcomes of Hematopoietic Cell Transplants from T-Replete Haploidentical Donors Using Post-Transplantation Cyclophosphamide with 10 of 10 HLA-A, -B, -C, -DRB1, and -DQB1 Allele-Matched Unrelated Donors and HLA-Identical Sibling Donors: A Multivariable Analysis Including Disease Risk Index. Biol Blood Marrow Transplant. 2016 Jan;22(1):125-33. doi: 10.1016/j.bbmt.2015.09.002. Epub 2015 Sep 7. PMID 26359881
- [Background] Ciurea SO, Mulanovich V, Saliba RM, Bayraktar UD, Jiang Y, Bassett R, Wang SA, Konopleva M, Fernandez-Vina M, Montes N, Bosque D, Chen J, Rondon G, Alatrash G, Alousi A, Bashir Q, Korbling M, Qazilbash M, Parmar S, Shpall E, Nieto Y, Hosing C, Kebriaei P, Khouri I, Popat U, de Lima M, Champlin RE. Improved early outcomes using a T cell replete graft compared with T cell depleted haploidentical hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2012 Dec;18(12):1835-44. doi: 10.1016/j.bbmt.2012.07.003. Epub 2012 Jul 11. PMID 22796535
- [Background] Raiola AM, Dominietto A, Ghiso A, Di Grazia C, Lamparelli T, Gualandi F, Bregante S, Van Lint MT, Geroldi S, Luchetti S, Ballerini F, Miglino M, Varaldo R, Bacigalupo A. Unmanipulated haploidentical bone marrow transplantation and posttransplantation cyclophosphamide for hematologic malignancies after myeloablative conditioning. Biol Blood Marrow Transplant. 2013 Jan;19(1):117-22. doi: 10.1016/j.bbmt.2012.08.014. Epub 2012 Aug 29. PMID 22940057
- [Background] Kanakry CG, Ganguly S, Zahurak M, Bolanos-Meade J, Thoburn C, Perkins B, Fuchs EJ, Jones RJ, Hess AD, Luznik L. Aldehyde dehydrogenase expression drives human regulatory T cell resistance to posttransplantation cyclophosphamide. Sci Transl Med. 2013 Nov 13;5(211):211ra157. doi: 10.1126/scitranslmed.3006960. PMID 24225944
- [Background] Ganguly S, Ross DB, Panoskaltsis-Mortari A, Kanakry CG, Blazar BR, Levy RB, Luznik L. Donor CD4+ Foxp3+ regulatory T cells are necessary for posttransplantation cyclophosphamide-mediated protection against GVHD in mice. Blood. 2014 Sep 25;124(13):2131-41. doi: 10.1182/blood-2013-10-525873. Epub 2014 Aug 18. PMID 25139358
- [Background] Stem Cell Trialists' Collaborative Group. Allogeneic peripheral blood stem-cell compared with bone marrow transplantation in the management of hematologic malignancies: an individual patient data meta-analysis of nine randomized trials. J Clin Oncol. 2005 Aug 1;23(22):5074-87. doi: 10.1200/JCO.2005.09.020. PMID 16051954
- [Background] Yang JZ, Zhang JQ, Sun LX. Mechanisms for T cell tolerance induced with granulocyte colony-stimulating factor. Mol Immunol. 2016 Feb;70:56-62. doi: 10.1016/j.molimm.2015.12.006. Epub 2015 Dec 17. PMID 26703218
- [Background] Jun HX, Jun CY, Yu ZX. In vivo induction of T-cell hyporesponsiveness and alteration of immunological cells of bone marrow grafts using granulocyte colony-stimulating factor. Haematologica. 2004 Dec;89(12):1517-24. PMID 15590404
- [Background] Deotare U, Al-Dawsari G, Couban S, Lipton JH. G-CSF-primed bone marrow as a source of stem cells for allografting: revisiting the concept. Bone Marrow Transplant. 2015 Sep;50(9):1150-6. doi: 10.1038/bmt.2015.80. Epub 2015 Apr 27. PMID 25915812
- [Background] Couban S, Messner HA, Andreou P, Egan B, Price S, Tinker L, Meharchand J, Forrest DL, Lipton J. Bone marrow mobilized with granulocyte colony-stimulating factor in related allogeneic transplant recipients: a study of 29 patients. Biol Blood Marrow Transplant. 2000;6(4A):422-7. doi: 10.1016/s1083-8791(00)70033-4. PMID 10975510
- [Background] Isola L, Scigliano E, Fruchtman S. Long-term follow-up after allogeneic granulocyte colony-stimulating factor--primed bone marrow transplantation. Biol Blood Marrow Transplant. 2000;6(4A):428-33. doi: 10.1016/s1083-8791(00)70034-6. PMID 10975511
- [Background] Ji SQ, Chen HR, Wang HX, Yan HM, Pan SP, Xun CQ. Comparison of outcome of allogeneic bone marrow transplantation with and without granulocyte colony-stimulating factor (lenograstim) donor-marrow priming in patients with chronic myelogenous leukemia. Biol Blood Marrow Transplant. 2002;8(5):261-7. doi: 10.1053/bbmt.2002.v8.pm12064363.
- [Background] Morton J, Hutchins C, Durrant S. Granulocyte-colony-stimulating factor (G-CSF)-primed allogeneic bone marrow: significantly less graft-versus-host disease and comparable engraftment to G-CSF-mobilized peripheral blood stem cells. Blood. 2001 Dec 1;98(12):3186-91. doi: 10.1182/blood.v98.12.3186. PMID 11719353
- [Background] Serody JS, Sparks SD, Lin Y, Capel EJ, Bigelow SH, Kirby SL, Gabriel DA, Wiley JM, Brecher ME, Schell MJ, Folds J, Shea TC. Comparison of granulocyte colony-stimulating factor (G-CSF)--mobilized peripheral blood progenitor cells and G-CSF--stimulated bone marrow as a source of stem cells in HLA-matched sibling transplantation. Biol Blood Marrow Transplant. 2000;6(4A):434-40. doi: 10.1016/s1083-8791(00)70035-8. PMID 10975512